CLINICAL TRIAL: NCT00857116
Title: The Impact of Deworming on Host Immunity and Clinical Outcome in Patients With Pulmonary Tuberculosis
Brief Title: Deworming Against Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: University of Gondar (Other); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Principal Investigator, Thomas Schon, MD PhD, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ALBP; HLF-20060245
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Tuberculosis
Keywords: Deworming; Tuberculosis; TB-score; Albendazole; Helminths
MeSH Terms: conditions — Tuberculosis | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albendazole (Active Comparator): Albendazole 400mg per os once daily for three consecutive days
  Interventions: Drug: Albendazole
- Placebo (Placebo Comparator): Placebo 400mg per os for three consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albendazole — Albendazole 400mg per os for three consecutive days at week 2 and week 8 after initiation of chemotherapy against tuberculosis
  Other Names: ALB
  Arms: Albendazole
Drug: Placebo — Placebo 400mg per os for three consecutive days at week 2 and week 8 after initiation of chemotherapy against tuberculosis
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether treatment against intestinal helminths in patients with pulmonary tuberculosis undergoing chemotherapy could improve the clinical outcome by enhancing host immunity.

DETAILED DESCRIPTION:
Mycobacterium tuberculosis causing tuberculosis (TB) is a major global public health problem. Because of increasing multi drug resistance and the long treatment period of at least six months, new therapeutic options are urgently needed. In countries like Ethiopia where TB is endemic, chronic worm infection is also highly prevalent. Recent data support that helminth infection might limit the host response against TB by inhibition of the TH1-response that is crucial in controlling the disease. In this study we want to test the hypothesis that Albendazole treatment of patients coinfected with helminths and TB could improve clinical outcome in addition to chemotherapy against TB. Additionally we will investigate the immunological interactions between TB and chronic helminths infection.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent to take part in the study
* Newly diagnosed pulmonary TB patients according to the WHO definitions of active tuberculosis who have a positive stool sample for helminths other than Schistosoma spp.

Exclusion Criteria:

* Pregnancy
* Corticosteroid or antibiotic treatment
* Symptomatic (diarrhoea) infection caused by worm infection
* Chronic diseases or acute infectious diseases other than TB or HIV
* Stool sample positive for Schistosoma spp

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-03; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in TB-score compared to baseline (Wejse et al 2007) | 2 months

SECONDARY OUTCOMES:
Sputum smear conversion | 3 months
Final outcome according to WHO | 6 months
Difference in ELIspot pattern (IL5, IFN-gamma and IL-10) | 3 months
Immunological response (IgE, Eosinophils, CD4-count) | 3 months
Chest X-ray improvement | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ebba Abate, MSc, Principal Investigator — University of Gondar and Linkoeping University; Ermias Diro, MD, Principal Investigator — University of Gondar; Thomas Schoen, MD PhD, Study Director — Linkoeping University, Sweden
Locations (1):
- University of Gondar, Gondar, Region 3, Ethiopia, Gondar, Ethiopia

REFERENCES:
- [Background] Borkow G, Bentwich Z. HIV and helminth co-infection: is deworming necessary? Parasite Immunol. 2006 Nov;28(11):605-12. doi: 10.1111/j.1365-3024.2006.00918.x. PMID 17042932
- [Background] Modjarrad K, Zulu I, Redden DT, Njobvu L, Lane HC, Bentwich Z, Vermund SH. Treatment of intestinal helminths does not reduce plasma concentrations of HIV-1 RNA in coinfected Zambian adults. J Infect Dis. 2005 Oct 1;192(7):1277-83. doi: 10.1086/444543. Epub 2005 Aug 25. PMID 16136473
- [Background] Kassu A, Mengistu G, Ayele B, Diro E, Mekonnen F, Ketema D, Moges F, Mesfin T, Getachew A, Ergicho B, Elias D, Wondmikun Y, Aseffa A, Ota F. HIV and intestinal parasites in adult TB patients in a teaching hospital in Northwest Ethiopia. Trop Doct. 2007 Oct;37(4):222-4. doi: 10.1258/004947507782333026. PMID 17988484
- [Background] Elias D, Akuffo H, Thors C, Pawlowski A, Britton S. Low dose chronic Schistosoma mansoni infection increases susceptibility to Mycobacterium bovis BCG infection in mice. Clin Exp Immunol. 2005 Mar;139(3):398-404. doi: 10.1111/j.1365-2249.2004.02719.x. PMID 15730384
- [Background] Elias D, Mengistu G, Akuffo H, Britton S. Are intestinal helminths risk factors for developing active tuberculosis? Trop Med Int Health. 2006 Apr;11(4):551-8. doi: 10.1111/j.1365-3156.2006.01578.x. PMID 16553939
- [Background] Elias D, Wolday D, Akuffo H, Petros B, Bronner U, Britton S. Effect of deworming on human T cell responses to mycobacterial antigens in helminth-exposed individuals before and after bacille Calmette-Guerin (BCG) vaccination. Clin Exp Immunol. 2001 Feb;123(2):219-25. doi: 10.1046/j.1365-2249.2001.01446.x. PMID 11207651
- [Derived] Abate E, Elias D, Getachew A, Alemu S, Diro E, Britton S, Aseffa A, Stendahl O, Schon T. Effects of albendazole on the clinical outcome and immunological responses in helminth co-infected tuberculosis patients: a double blind randomised clinical trial. Int J Parasitol. 2015 Feb;45(2-3):133-40. doi: 10.1016/j.ijpara.2014.09.006. Epub 2014 Dec 5. PMID 25486494